CLINICAL TRIAL: NCT04405791
Title: Efficacy of Clinical Application of Transcranial Low Intensity Focused Ultrasonic Stimulation for Patients With Major Deperessive Disorder - Exploratory Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Ho Seok, Professor, Department of Psychiatry, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3-2018-0352
Record Dates: First submitted 2020-05-21; First posted 2020-05-28 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Major Depressive Disorder(MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Clinical psychologists who participate in diagnosis and symptom evaluation and subjects conduct double-blindness that make it impossible to know which group they are assigned to, and only the PI and treatment implementer can know the allocation group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation group (Experimental): "low intensity transcranial focused ultrasound (tFUS) stimulation"The acoustic intensity output of the FUS transducer was validated at the maximum intensity area using a calibrated needle hydrophone (HNR-500, Onda). The incident acoustic intensity and pressure at the FUS focus were 3W/cm2 spatial-peak pulse-average acoustic intensity (Isppa) and a peak negative pressure (Pr) of 300 kPa. The incident acoustic intensity and pressure at the FUS focus were 3W/cm2, and tone burst duration was 1 ms at 50 % duty cycle (thus, pulse repletion frequency was 500 Hz) for the duration of 300 ms, according to the studies in humans. Each sonication was delivered every 6 s for the duration of 20 min (a total FUS stimulation per each session was therefore 200 times). With a derating factor of 55% reduction in pressure transmission by the human skull, estimated in situ Pr was ~135 kPa with an in situ acoustic intensity of 600 mW/cm2 Isppa .
  Interventions: Procedure: Active stimulation group Sham stimluation group
- Sham stimluation group (Sham Comparator): "sham stimulation" In case of sham stimulation, the same procedure was repeated without providing actual sonication. No subjects in FUS condition hear/feel any tangible somatosensory phenomena; therefore, the sham condition was indistinguishable.
  Interventions: Procedure: Active stimulation group Sham stimluation group

INTERVENTIONS:
Procedure: Active stimulation group Sham stimluation group — Participants are randomly assigned to either treatment group or sham group for application of transcranial low intensity focused ultrasound stimulation. For sham group, transducer is surrounded by rubber band in order to block the transmission of ultrasonic wave.
  Before initiating transcranial low intensity focused ultrasonic stimulation, in order to identify anatomical structure of the brain, Brain Magnetic Resonance Image(MRI) and Computer Tomography(CT) will be taken. For image coordination, multi-modal stick(fiducial marker, PinPoint) will be attached to the participant.
  With acquired brain images of the participant, researchers identify participant's dorsolateral prefrontal cortex(DLPFC) region, and design focused ultrasound focus targeting, image-guidance method.
  The treatment is started by targeting left DLPFC region according to assigned groups. Both the treatment and sham group will be under procedure for 2 weeks, 3 times a week.

SUMMARY:
The non-invasive type ultrasonography system is applied to patients with major depressive disorder to evaluate their effectiveness and safety. Brain Computer Tomography(CT) and Magnetic Resonance Image(MRI) are taken to induce images before transcranial low intensity focused ultrasonic stimulation.

Through random extraction, the group is divided into treatment group and placebo group. The treatment is started by targeting left Dorsolateral prefrontal cortex(DLPFC) region according to assigned groups. As for women, considering mood change during menstrual cycle, the treatment is taken place 1 week after the menstruation has initiated. The treatment group and the placebo group will be treated three times a week for two weeks.

To evaluate clinical symptoms, Quick Inventory of Depressive Symptomatology-Self Report, Scale for Suicidal Ideation, state-trait anxiety scale, frontal lobe management function test, memory test, and continuous performance test are performed before, during, and after treatment. For the assessment of side effects, Systematic Asseseement for Treatment Emergent Events-General Inquiry(SAFTEE) are conducted for treatment presentation events every week during the treatment implementation period and every two weeks after the treatment is completed.

ELIGIBILITY:
Inclusion Criteria:

1)19 to 60 years of age 2)Having major depressive disorder without psychotic feature according to the DSM-5 diagnosis criteria SCID-5-CV: (ICD-10 code : F32.0, F32.1, F32.2, F33.0, F33.1, F33.2) 3)Montgomery-Asberg Depression Rating Scale (MADRS) score ≥12 4)No history of suicidal attempt with suicidal ideation tendency score assessed by the Scale for Suicide Ideation (SSI) ≤ 9 5)No antidepressants regimen for 4 weeks prior to enrollment. 6)n the case of active antidepressants regimen, patients with MADRS score ≥12 and who will not change their medication doses during the study period

Exclusion Criteria:

* Incompatibility with brain CT and MRI
* Disorders that may cause depression (e.g., thyroid dysfunction, uncontrolled diabetes) or who taking medications that can influence on mood (e.g., thyroid hormones, steroids.)
* History of epileptic seizures
* History of major psychiatric disorder including schizophrenia and bipolar disorder
* Mental retardation
* Severe physical illness including cancer and tuberculosis
* Significant skin problems including contact dermatitis
* Pregnant women or women planning to become pregnant
* (After CT scan) skull thickness ≥ 8, or significant calcification
* (After MRI scan) structural abnormalities such as brain tumors, hemorrhage, traumatic brain disease, or structural changes due to degenerative brain disorders

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Change in Montogmery-Asberg Depression Rating Scale, MADRS | 1. Baseline assessment (pre-intervention: active or sham)2. Second assessment (Immediately after the active or sham stimulation) 3.Third assessment(Two weeks after the active or sham stimulation)
  MADRS is a clinician rating scale for depression

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, Gangnam, South Korea